CLINICAL TRIAL: NCT00166634
Title: The Role of Ambulatory Blood Pressure Monitoring (ABPM) in Interventional Trials Conducted in Children With Hypertension
Brief Title: Ambulatory Blood Pressure Monitoring in Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Pediatric Pharmacology Research Units Network (Network)
Responsible Party: Leah Dawson, Arkansas Children's Hospital Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PPRU 10668s
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Hypertension
Keywords: Hypertension; ABPM; Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ambulatory Blood Pressure Monitoring (ABPM)

SUMMARY:
The primary objective of this proposal is to demonstrate that ABPM can be used to improve study design for interventional trials in children with hypertension.

DETAILED DESCRIPTION:
ABPM is a standard technique in adult antihypertensive trials to study the magnitude and duration of effect of investigational drugs. These methods are needed for pediatric studies. Before such methods can be developed, preliminary information must be collected to demonstrate that the device can be used for antihypertensive studies in children (i.e, to determine the dropout rate following the first ABP study, to determine the frequency of white coat hypertension in a selected population, to compare casual (office) blood pressures commonly used to diagnose hypertension in children with those obtained by ABPM, and to assess the placebo effect in children with borderline and mild hypertension).

All participants will be asked to complete 24 hour ABPM on two occasions within one week. During the ABPM parents and children will be asked to keep a diary recording the times that the child slept. A crossover design will be used, where subjects are initially randomized to either drug or placebo and then will be crossed over to the other intervention at a set time during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children 5-16 years of age.
* Borderline or mild systolic and or diastolic hypertension as defined by 1996 Task Force criteria.
* No current drug therapy for hypertension being taken.
* Must be ambulatory and willing to wear an ABP monitor for 24 hours
* Agree to refrain from swimming, showering and other activities that might result in damage to ABP monitor during the two 24 hour intervals that the monitor is worn.
* Standing height between 45 inches and 73 inches
* Informed parental consent and patient assent.

Exclusion Criteria:

* Severe or life threatening hypertension.
* Any drug therapy that may raise or lower the blood pressure.
* Any severe bleeding disorder or concurrent treatment with anticoagulant medications
* Non-ambulatory
* Significant arrhythmia
* Previous history of significant non-compliance with prescribed medical care.
* Any other disease that, in the opinion of the investigator, might interfere with the accurate measurement of the blood pressure or place the subject at risk unnecessarily.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2003-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is ABPM to examine borderline high blood pressure, mild or untreated blood pressure in children captured within a 24 hour period on two occasions within a week.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kosair Children's Hospital, Louisville, Kentucky
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Utah--Primary Children's Medical Center, Salt Lake City, Utah